CLINICAL TRIAL: NCT05676385
Title: Glucose Response to a Formula for Patients at Risk of Hypoglycaemia
Acronym: EFFECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SBB22R&52507
Record Dates: First submitted 2022-12-12; First posted 2023-01-09 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Postprandial Hypoglycemia
Keywords: nutritional product; glucose response; carbohydrate metabolism
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Intervention Model Description: Randomised, controlled, double-blind, cross-over, single-centre, Proof of-Concept study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dietary supplement/First concept Product 1 (containing 50 grams of carbohydrates) (Active Comparator): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: First concept product (containing 50 grams of carbohydrates); Dietary Supplement: Second concept product (containing 50 grams of carbohydrates); Dietary Supplement: Reference product (containing 50 grams of carbohydrates)
- Dietary supplement/First concept Product 2 (containing 50 grams of carbohydrates) (Active Comparator): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized
  Interventions: Dietary Supplement: First concept product (containing 50 grams of carbohydrates); Dietary Supplement: Second concept product (containing 50 grams of carbohydrates); Dietary Supplement: Reference product (containing 50 grams of carbohydrates)
- Reference product (containing 50 grams of carbohydrates) (Active Comparator): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized
  Interventions: Dietary Supplement: First concept product (containing 50 grams of carbohydrates); Dietary Supplement: Second concept product (containing 50 grams of carbohydrates); Dietary Supplement: Reference product (containing 50 grams of carbohydrates)

INTERVENTIONS:
Dietary Supplement: First concept product (containing 50 grams of carbohydrates) — Fasted intake of First concept product (randomised)
Dietary Supplement: Second concept product (containing 50 grams of carbohydrates) — Fasted intake Second concept product (randomised)
Dietary Supplement: Reference product (containing 50 grams of carbohydrates) — Fasted intake of Reference product (randomised)

SUMMARY:
This study assesses the glycemic responses to several nutritional products.

DETAILED DESCRIPTION:
During a study visit fasted subjects will consume one serving of the reference product or of the test products. Venous blood samples will be taken at baseline and at several time-points over a 6-hr period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals, 18 up to and including 50 years of age.
2. Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial.
3. Willing to avoid the consumption of alcohol, unusual food intake, unusual physical activity 24h prior to each study visit.
4. Willing to come to the study visit in the morning after an overnight fast of minimum 10 hours and maximum 14 hours (with water only).

Exclusion Criteria:

1. Blood glucose levels ≥ 7.8 mmol/L at screening (not fasted)
2. Known history of gastrointestinal disease (e.g., diverticulitis, Crohn's disease, coeliac disease etc.), bariatric surgery, AIDS, hepatitis, a history or presence of clinically important endocrine (including Type 1 or Type 2 diabetes mellitus), or any condition which might, in the opinion of the Principal Investigator either: 1) make participation dangerous to the subject (e.g. anaemia) or to others, or 2) affect the results.
3. Use of medications known to influence carbohydrate metabolism, gastrointestinal function or appetite, including, but not limited to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids within 4 weeks of the screening visit, or any medication which might, in the opinion of the Principal Investigator either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
4. Use of medications known to influence gastric emptying (including but not limited to anticholinergics, nicotine, narcotic analgesics, ganglion blocking drugs, antacids and metoclopramide).
5. Use of anti-clotting medications.
6. Current tobacco smokers or smokers that quite smoking < 1 month prior to screening (except for occasional (≤ 3) cigarettes/cigars/pipes per week on average over the past month).
7. Self-reported pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Decline in glucose level after reaching peak (Cmax) | 6 hours
  The decline in glucose (mmol/hour) after reaching peak glucose levels (Cmax) until reaching baseline (t = -5) blood glucose levels or, in case baseline blood glucose levels are not reached, the lowest observed blood glucose level.

SECONDARY OUTCOMES:
Incremental Area Under the Curve (iAUC) for glucose | 6 hours
  Incremental Area Under the Curve (iAUC) for glucose (mmol/L/hrs)
Incremental Area Under the Curve (iAUC) for insulin | 6 hours
  Incremental Area Under the Curve (iAUC) for insulin (pmol/L/hrs)
Incremental Area Under the Curve (iAUC) for paracetamol | 6 hours
  Incremental Area Under the Curve (iAUC) for paracetamol (pmol/L/hrs)
Incremental peak levels (iCmax) of glucose | 6 hours
  Incremental peak levels (iCmax) of glucose (mmol/L)
Incremental peak levels (iCmax) of insulin | 6 hours
  Incremental peak levels (iCmax) of insulin (pmol/L)
Incremental peak levels (iCmax) of paracetamol | 6 hours
  Incremental peak levels (iCmax) of paracetamol (mg/L)
Time to peak levels (Tmax) of glucose | 6 hours
  Time to peak levels (Tmax) of glucose (min)
Time to peak levels (Tmax) of insulin | 6 hours
  Time to peak levels (Tmax) of insulin (min)
Time to peak levels (Tmax) of paracetamol | 6 hours
  Time to peak levels (Tmax) of paracetamol (min)

CONTACTS AND LOCATIONS:
Locations (1):
- EB UtrechtResearch BV, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No